CLINICAL TRIAL: NCT00963521
Title: Pilot Study of Therapeutic Vaccination by Leukemic Blasts in Vitro Differentiated Dendritic Cells From Patients With Acute Myelogenous Leukemia in Complete Remission
Brief Title: Vaccine Therapy in Treating Patients With Acute Myeloid Leukemia in Complete Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000626786; IPC-2006-011; INCA-RECF-0628; EUDRACT-2006-007093-29; IPC-LADC
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Leukemia
Keywords: adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Congenital Abnormalities

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from dendritic cells may help the body build an effective immune response to kill cancer cells.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy and to see how well it works in treating patients with acute myeloid leukemia in complete remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the tolerability of autologous dendritic cell vaccine in patients with acute myelogenous leukemia in complete remission.

Secondary

* Evaluate the emergence of an immune response.
* Determine the relapse rate.
* Assess the occurrence of residual disease.

OUTLINE: Patients receive increasing doses of blastic cells transformed in vitro by autologous dendritic cells (1/3 subcutaneously and 2/3 IV) every 3 weeks for up to 5 doses.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myelogenous leukemia (AML)

  * Myelomonocytic (M4) or monocytic (M5) subtype
  * In second complete remission (CR) or later following CR1 lasting ≤ 12 months after chemotherapy that may have included an intensification regimen followed by autologous transplantation
* No (15;17) translocation
* No AML M3
* HLA-A2 positivity
* CD14 ≥ 20% on peripheral blood mononuclear cells
* Circulating blasts ≥ 10 x 109/L (collected prior to chemotherapy) available
* Must not be eligible for HLA-matched allogeneic transplantation
* No progressive disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No contraindication to cytopheresis or chemotherapy
* No HIV or HTLV positivity
* No hepatitis B or C activation
* No prior psychological disease
* Not deprived of liberty and able to give consent
* Must be able to speak and read French
* No other cancer except for basal cell or cervical

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent participation in another clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Adverse events at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Chabannon, MD, PhD — Institut Paoli-Calmettes
Locations (1):
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France